CLINICAL TRIAL: NCT02335177
Title: Technology and Human Help at Home After Hospitalisation (T4H): a Randomized Clustered Controlled Trial
Brief Title: Technology and Human Help at Home After Hospitalisation
Acronym: T4H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ages et Vies Association (Other)
Collaborators: Caisse Nationale de Solidarité pour l'Autonomie (Other); National Insurance Fund Vieilleisse (Other); Réunica (Unknown); Fondation Macif (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-A00579-38
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Patient Fall
Keywords: Falls; Elderly; Physical activities; Technologies for autonomy; Impact of intervention; autonomy; physical activity program
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventionnal arm (Active Comparator): Interventional arm : patients at home with technologies for autonomy and tailored physical activity program.
  Interventions: Behavioral: Interventional arm
- Control arm (No Intervention): Control arm : patients with usual care home

INTERVENTIONS:
Behavioral: Interventional arm — At home patients have both technologies for autonomy (walkers, treadmill) and tailored physical activity program performed with the help of the home carer. Intervention takes 3 months. Assessment at hospital discharge et at 3 months.
  Arms: Interventionnal arm

SUMMARY:
Elderly people are still at risk for falling at home. The objective of the study is to evaluate at home the impact of an intervention for 3 months combining technologies for autonomy and tailored physical activity program. The study is performed among patients aged 75 years and over leaving Charles Foix Geriatrics hospital or already supported by carer of professional home-care service Ages & Vie and with a loss of autonomy requiring physiotherapy and home support workers. It is a prospective, randomized, single-center, in cluster study which compares a Patient group (interventional group) with the intervention program (technologies + physical activities) with a control group benefiting from usual care home. Our hypothesis is that in the interventional group fewer falls were observed and improved different scores (Timed Up and Go Test,Barthel index, Quality of Life questionnaire of Duke) were reported compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in Charles Foix Hospital (France) and returning home or already supported by carer of professional home-care service Ages & Vie
* > 75 years old with loss of autonomy
* at risk for falling
* able to read and understand the information letter and consent letter
* patient requiring physiotherapy and caregiver at home.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of falls | 3 months
  absence of fall requiring medical or paramedical care and improvement of the Timed Up and Go Test (TUG) or improvement of the autonomy level assessed by Barthel Index with at least stability of the test that is not improved

SECONDARY OUTCOMES:
Timed up and Go test score | 3 months
Barthel index | 3 months
Duke questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Meziere Anthony, Dr, Principal Investigator — Hôpital Charles Foix, AP-HP
Locations (1):
- AP-HP Charles Foix, Ivry-sur-Seine, France

REFERENCES:
- [Derived] Meziere A, Oubaya N, Michel-Pellegrino V, Boudin B, Neau M, Robert H, Cara I, Salgado Sanchez L, Baloul S, Piette F, Pautas E, Picou Y, Curtis V, Schonheit C, Canoui-Poitrine F, Moreau C. Exercise Interventions With Trained Home Helpers for Preventing Loss of Autonomy and Falls in Community-Dwelling Older Adults Receiving Home Heath Physical Therapy T4H: A Randomized Controlled Pilot Study. J Geriatr Phys Ther. 2021 Jul-Sep 01;44(3):E138-E149. doi: 10.1519/JPT.0000000000000287. PMID 33534333